CLINICAL TRIAL: NCT06056115
Title: Efficacy and Safety of Tislelizumab Combined With Platinum-containing Drug Chemotherapy in First-line Treatment of Lung Adenocarcinoma With Asymptomatic Brain Metastatic
Brief Title: Efficacy and Safety of Tislelizumab for Lung Adenocarcinoma With Asymptomatic Brain Metastatic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jian SHI, Professor, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220511
Record Dates: First submitted 2023-04-11; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — tislelizumab; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab Combined With Platinum-containing Drug Chemotherapy (Experimental): 1. Tislelizumab PD-1 inhibitor
  2. Platinum-containing drug chemotherapy
  Interventions: Drug: Tislelizumab,Platinum

INTERVENTIONS:
Drug: Tislelizumab,Platinum — 1. Induction therapy stage:
     Tislelizumab plus platinum-containing drug chemotherapy was administered every 3 weeks and was expected to complete 6 cycles of treatment.
  2. Maintenance treatment phase:
  After completion of the induction therapy phase, patients whose antitumor response was confirmed as complete response, partial response, and disease stable according to RECIST v1.1 criteria were admitted to maintenance therapy .

SUMMARY:
Brain metastasis of lung cancer is one of the most important metastasis pathways in patients with life-threatening diseases. This study explore the efficacy and safety of Tislelizumab combining with platinum-containing drug chemotherapy in the first-line treatment of Lung Adenocarcinoma With Asymptomatic Brain Metastatic. Meanwhile, Related biomarkers were explored to provide theoretical basis for efficacy evaluation and resistance mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic (stage IV) lung adenocarcinoma who have not been systematically treated and are histologically or cytologically confirmed as unable to undergo radical surgery or radiotherapy based on AJCC Stage VIII;
2. Patients with brain metastases confirmed by imaging;
3. Patients with asymptomatic BMS after initial diagnosis, local BMS surgery or radiotherapy;
4. ECOG PS: 0-1;
5. Measurable target lesions outside the skull (as per RECIST 1.1);
6. Life expectancy greater than 3 months;

Exclusion Criteria:

1. Patients had been treated with immune checkpoint inhibitors such as anti-PD-1, PD-L1, or CTLA-4 therapy;
2. The patient had received systemic chemotherapy as advanced treatment;
3. Patients with EGFR mutation or ALK gene translocation;
4. The patient had received approved systemic anticancer therapy or systemic immunomodulators (including but not limited to interferon, interleukin 2, and tumor necrosis factor) within 4 weeks prior to initial administration;
5. Clinically uncontrolled pleural fluid or ascites requiring puncture drainage within 2 weeks prior to initial administration;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
1 years PFS | up to 1year
  the time from the date of first dose of study treatment to the date of first documentation of disease progression using RECIST v1.1 or death, whichever occurs first

SECONDARY OUTCOMES:
The objective response rate (ORR) | Through study completion, an average of 12 months
  Assessed by the Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jian Shi, Dr., Principal Investigator — The Fourth Hospital of Hebei Medical University (Hebei Tumor Hospital)
Locations (1):
- The Fourth Hospital of Hebei Medical University (Hebei Tumor Hospital), Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No